CLINICAL TRIAL: NCT05841069
Title: Multicenter Controlled Randomized Prospective Study of the Comparative Efficacy of Early and Delayed Surgical Interventions in Patients With Acute Adhesive Intestinal Obstruction
Brief Title: Short and Prolonged Conservative Treatment in Patients With Adhesive Intestinal Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: North-Western State Medical University named after I.I.Mechnikov (Other)
Responsible Party: Principal Investigator, Kotkov Pavel, PhD, surgery department assistant, North-Western State Medical University named after I.I.Mechnikov
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24121989
Record Dates: First submitted 2023-04-11; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Small Bowel Obstruction; Small Bowel Adhesion
Keywords: Acute adhesive intestinal obstruction, conservative treatment
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Intervention Model Description: Multicenter controlled randomized prospective study
Masking Description: No masking is expected due to the nature of interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short conservative treatment (Active Comparator): Conservative treatment will be performed within no more than 24 h. Surgery will be performed in the absence of contrast in colon according to X-ray examination and if signs of clinical degradation will appear.
  Interventions: Procedure: Adhesiolysis; Radiation: X-ray examination; Procedure: Conservative treatment
- Prolonged conservative treatment (Experimental): Conservative treatment will be performed within N h, where N = 72 h minus duration of acute intestinal obstruction. Surgery will be performed in the absence of contrast in colon according to X-ray examination and if signs of clinical degradation will appear.
  Interventions: Procedure: Adhesiolysis; Radiation: X-ray examination; Procedure: Conservative treatment

INTERVENTIONS:
Procedure: Adhesiolysis — Median laparotomy with subsequent detection of intestinal obstruction cause and adhesiolysis.
Radiation: X-ray examination — Plain X-ray of abdomen (1-4 times) with water insoluble contrast.
Procedure: Conservative treatment — A set of measures aimed at non-operative resolution of acute intestinal obstruction - nasogastric tube, infusion therapy.

SUMMARY:
This study will compare the results of 24 h conservative treatment and N h conservative treatment of adhesive small bowel obstruction (where N = 72 h minus duration of intestinal obstruction).

DETAILED DESCRIPTION:
Patients with acute adhesive intestinal obstruction, who dont need an emergency operation, will be given water insoluble contrast per os and randomized into two groups - early and delayed surgery. The first group will receive conservative treatment within no more than 24 h. Duration of non-operative treatment in second group will be 72 h minus duration of intestinal obstruction, based on the onset of symptoms. In both groups surgery will be performed if contrast will not reach colon in mentioned terms or clinical deterioration signs will appear. The results of 24 h conservative treatment and N h conservative treatment (where N = 72 h minus duration of intestinal obstruction) will be compared.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute intestinal obstruction

Exclusion Criteria:

* pregnancy;
* peritonitis or strangulation, revealed during primary examination;
* early acute small bowel obstruction (presence of anamnestic surgical intervention within 6 month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Non-operative treatment success | 72 hours
  Frequency of non-operative intestinal obstruction resolution

SECONDARY OUTCOMES:
Overall mortality | up to 30 days
  Number of patients, died during hospitalization
Postoperative complications | up to 30 days
  Number and variety of postoperative complications in patients, who underwent surgery
Resectional interventions | up to 30 days
  Number of patients, who underwent surgery, including small bowel resection

CONTACTS AND LOCATIONS:
Locations (4):
- Russia (4):
  - 26 City Hospital, Saint Petersburg
  - North-Western State Medical University named after I. I. Mechnikov, Saint Petersburg
  - Saint-Petersburg I.I. Dzhanelidze Research Institute of Emergency Medicine, Saint Petersburg
  - The City Hospital of the Holy Martyr Elizabeth, Saint Petersburg

IPD SHARING:
Plan to Share IPD: Undecided